CLINICAL TRIAL: NCT04322825
Title: Mollii - Personalized Suit for Treatment of Spasticity, GFMCS3-5
Brief Title: Mollii - Personalized Suit for Treatment of Spasticity, GFMCS 3-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Eurostars (Other)
Responsible Party: Principal Investigator, christian wong, principle investigator, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-17004467
Record Dates: First submitted 2019-11-01; First posted 2020-03-26 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Spastic Cerebral Palsy
Keywords: Mollii suit;; Goal Attainment Scale;; Reciprocal inhibition;; modified ashworth scale,; trans cutaneous electric stimulation, TENS; Spasticity reduction,
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): 24 weeks of TENS
  Interventions: Device: TENS incorporated into the Mollii suit

INTERVENTIONS:
Device: TENS incorporated into the Mollii suit — trans cutaneous electric stimulation,

SUMMARY:
The objective of this study was to examine the effect on spasticity and function of multifocal transcutaneous electrical stimulation incorporated in a 2-piece (Mollii) suit.

DETAILED DESCRIPTION:
In this prospective cohort study, the participants (children with predominantly spastic CP, GFMCS 3-5) wore the suit for 1 hour every second day for 24 weeks. The investigators evaluated level of spasticity using the modified Ashworth scale (MAS) and other related measures before initiation, after 4, 12, and 24 weeks. Two motor related smart goals were defined and evaluated by the goal attainment scale (GAS). GMFM-66 and posture and postural ability scale (PPAS) were performed.

ELIGIBILITY:
Inclusion Criteria:

- cerebral palsy with spastic disease, GMFCS 3-5.

Exclusion Criteria:

* other disorders affecting the sensorimotor functions without spasticity,
* implanted electric medical devices,
* BMI>35
* other severe concomitant diseases such as cancer, cardiovascular, inflammatory, psychiatric disease, medical dysregulated epilepsy or hypertension.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
modified ashworth scale | 24 weeks
  spasticity evaluation from 0 (best) to 4 (worst) in modified ashworth scale

SECONDARY OUTCOMES:
Goal Attainment Scale | 24 weeks
  smart goals from -2 (worst) to +2 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- hospital of Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
we are not permitted to share these data due to gpdr ruels